CLINICAL TRIAL: NCT06579326
Title: Multistructural Quantitative Photoacoustic Imaging of Human Feet With Lower Extremity Artery Disease
Brief Title: Photoacoustic Tomography in Assessment of Lower Extremity Artery Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jia Liu, Principal Investigator, Sun Yat-sen University
Other Study IDs: II2024-189-02
Record Dates: First submitted 2024-08-27; First posted 2024-08-30 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Lower Extremity; Photoacoustic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Photoacoustic imaging — It could provide three-dimensional ultrasound images of vessels in the target area. It could also provides super-resolution and large-depth photoacoustic images. By effectively extracting photoacoustic spectral features and using spectral feature unmixing algorithm, blood oxygen saturation can be calculated.

SUMMARY:
Lower extremity artery disease (LEAD) is characterized by low awareness rate and high missed diagnosis rate, leading to low treatment rate and high disabling mortality rate. However, none of the current examination methods can comprehensively and thoroughly evaluate the vascular structure and blood oxygen status of the lower extremity at the same time. Photoacoustic imaging can display millimeter-scale microvessels without the need for contrast agents. The investigators developed photoacoustic tomography (PACT) technology, which wass able to provide three-dimensional and high-resolution photoacoustic images of the target area.The investigators plan to recruit LEAD patients in different disease conditions and healthy volunteers to receive the PACT examination on the feet using this imaging system, and to evaluate the potential clinical role of the imaging system in LEAD, and its added value to current imaging methods.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion of the case group 1) LEAD patients; 2) Patients voluntarily take part in the study and write informed consent.
2. Inclusion of the control group 1) Patients without LEAD by ultrasound and clinical diagnosis; 2) Patients voluntarily take part in the study and write informed consent.

Exclusion Criteria:

1. age <18 years;
2. pregnant women, nursing mothers and pregnant women in preparation;
3. with laser operation contraindication (for example, received a photodynamic therapy in the last month);
4. with metal implants in lower legs or feet;
5. with a history of mental illnesses or abuse of drug and alcohol;

7) with blood phobia or pathological hypotension; 8) with cerebral hemorrhage or peripheral vascular bleeding risk, or history of stroke; 9) with wounds in lower legs or feet; 10) unable or uncooperative with the experimenter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The LEAD patients are diagnosed as LEAD by computed tomography angiography or ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean vessel density of foot vasculature measured by photoacoustic imaging | Baseline
  Vessel density (number of vessels per mm²) in foot vasculature will be quantified using photoacoustic imaging. Results will be reported as mean ± SD.

SECONDARY OUTCOMES:
Mean oxygen saturation in pedal vasculature measured by photoacoustic imaging | Baseline
  Oxygen saturation in pedal vasculature will be quantified by photoacoustic imaging. Results will be reported as mean ± SD. Unit of Measure: %
Mean hemoglobin concentration in pedal vasculature measured by photoacoustic imaging | Baseline
  Description: Hemoglobin concentration in pedal vasculature will be quantified by photoacoustic imaging. Results will be reported as mean ± SD.
  Unit of Measure: g/dL

CONTACTS AND LOCATIONS:
Locations (1):
- the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China